CLINICAL TRIAL: NCT01859442
Title: Phase 1 Study of Mitochondrial Energetics After Long Course Chemoradiotherapy and a Short Term Exercise Programme in Locally Advanced Rectal Cancer Patients - A Randomized Controlled Trial.
Brief Title: The Effect of Cancer Therapies and Exercise on Mitochondrial Energetics and Fitness
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michelle Mossa (Other Government)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor-Investigator, Michelle Mossa, Research an Developement Deputy Director, Liverpool University Hospitals NHS Foundation Trust
Organization: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11/H1002/12c
Record Dates: First submitted 2013-05-13; First posted 2013-05-22 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2013-09

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Active Comparator): 6 week structured responsive interval exercise training programme
  Interventions: Procedure: Structured responsive interval exercise training programme
- Control group (Sham Comparator): Negative, unsupervised, out of hospital control group
  Interventions: Other: Sham group

INTERVENTIONS:
Procedure: Structured responsive interval exercise training programme
  Arms: Exercise group
Other: Sham group — NO intervention in this group, only standard care (no exercise programme)
  Arms: Control group

SUMMARY:
The present study is a randomised control trial investigating the effects of a short six week exercise training program in rectal cancer patients following neoadjuvant chemoradiotherapy prior to elective rectal cancer surgery.

Twelve patients will be randomised (1:1) to an intervention and a control group. The patients randomized to the intervention group will attend a total of 18 tailored exercise sessions (Three 40 minute sessions for six weeks) after their 6 weeks of chemoradiotherapy treatment. Where possible the exercise training sessions will be arranged to fit in with other appointments at the hospital. Patients randomized to the control group will be unsupervised. They will only attend an extra 3 sessions were a cardiopulmonary exercise test and VO2 Kinetics test will be performed. Patients will also be invited to attend 3 health related quality of life interviews at week 0, 3 and 6 during their exercise programme. These appointments will be directly before or after their exercise sessions to minimise hospital attendence.

Following surgery only routine clinically relevant observational data will be collected. These data will relate to hospital length of stay, the level of care required following surgery, post-operative morbidity survey (POMS) and the recovery process. Most of this information can be accessed from patient notes and on the electronic patient records system.

This is a subgroup RCT of patients in a larger interventional trial (6 control and 6 exercise intervention patients) will be asked to consent separately for the the 31-Phosphorus Magnetic Resonance Spectroscopy (31P MRS) scans and the blood samples.

HYPOTHESIS

1. Interval exercise training will maintain or improve fitness (measured by anaerobic threshold) in patients undergoing neoadjuvant chemoradiotherapy.
2. Interval exercise training is safe and feasible in patients undergoing neoadjuvant chemoradiotherapy awaiting rectal cancer resection.
3. Interval exercise training will improve other measures of physical fitness measured in the CPET and the oxygen uptake kinetics test.
4. Interval exercise training will improve quality of life in patients undergoing neoadjuvant chemoradiotherapy.
5. Improvements in physical fitness will reduce postoperative complications following major rectal cancer surgery.
6. Does physical activity, measured by Sensewear Pro 3 activity monitors, decrease during neoadjuvant chemoradiotherapy and can this decrease be attenuated by an exercise training program?
7. Can we find an optimal time for surgery when fitness and cancer downstaging are at their best?

HYPOTHESIS for Mechanism Pilot Study

1. To explore the exponential rate constant of post-exercise phosphocreatine recovery.
2. To explore the alteration in cellular and mitochondrial energetics eg. Change in mitochondrial numbers, change in mitochondrial activity and respiration.

DETAILED DESCRIPTION:
All patients will attend 5 sets of appointments at the hospital for diagnostic tests and 3 appointments at the University of Liverpool Magnetic Resonance and Image Analysis Research Centre (MARIARC). Three appointments will be prior to chemoradiotherapy treatment, and the other 4 will be after chemoradiotherapy. Two of these 5 appointments are part of routine care. The first 4 appointments will last about an hour. Patients will complete 3 quality of life questionnaires on recruitment, during chemotherapy, before and 4-6 weeks after surgery. These 3 questionnaires will take 20 minutes to fill in. The fourth and fifth appointments will consist of Computed Tomogram (CT) and Magnetic Resonance Imaging (MRI) scans in our radiology department to assess cancer staging. These appointments will last about 1 hour 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of T3N+ rectal cancer
* above age of 18
* able to conduct a cardiopulmonary exercise test on a cycle ergometer

Exclusion Criteria:

* unable to conduct a cardiopulmonary exercise test on a cycle ergometer
* metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Exponential rate constant of post-chemoradiotherapy and post-exercise phosphocreatine recovery. | Between baseline and week 0 and between week 0 at week 6 post-NACRT

SECONDARY OUTCOMES:
Alterations in mitochondrial energetics post-chemoradiotherapy and exercise | Between baseline and week 0 and between week 0 and week 6 post-NACRT
  Changes in 31- Phosphoromagnetic resonance spectroscopic (31-PMRS) ATP:ADP ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Aintree University Teaching Hospitals NHS FT, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] West MA, Loughney L, Lythgoe D, Barben CP, Adams VL, Bimson WE, Grocott MP, Jack S, Kemp GJ. The effect of neoadjuvant chemoradiotherapy on whole-body physical fitness and skeletal muscle mitochondrial oxidative phosphorylation in vivo in locally advanced rectal cancer patients--an observational pilot study. PLoS One. 2014 Dec 5;9(12):e111526. doi: 10.1371/journal.pone.0111526. eCollection 2014. PMID 25478898